CLINICAL TRIAL: NCT06825507
Title: Stepped Care Model of Lifestyle-based Mental Health Care for Depression: a Randomised Controlled Trial and Economic Evaluation
Brief Title: Stepped Care Model of Lifestyle-based Mental Health Care for Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assoicate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY036
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Depression
Keywords: Stepped care model; Lifestyle medicine; Randomised controlled trial; Cost-effectiveness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle-based mental health care (LSC) (Experimental): Participants in the LSC will access a 6-month lifestyle-based stepped care treatment for depression.
  Interventions: Behavioral: Lifestyle-based mental health care
- Care-as-usual (CAU) (Other): Participants in the CAU will have unrestricted access to mental health services based on their needs and preferences.
  Interventions: Other: Care-as-usual

INTERVENTIONS:
Behavioral: Lifestyle-based mental health care — Participants in the LSC will access a stepped care treatment consisting of 3 steps, including self-help multicomponent LM treatment (Step 1), guided self-help based on the LM approach and low-intensity cognitive behavioural therapy for depression (Step 2), and specialist mental health services (Step 3).
  Arms: Lifestyle-based mental health care (LSC)
Other: Care-as-usual — Participants in the CAU will receive their baseline depressive symptom severity via text message following randomisation, and they will have unrestricted access to mental health services based on their needs and preferences, such as pharmacological treatments, psychological treatments, and complementary and alternative medicine.
  Arms: Care-as-usual (CAU)

SUMMARY:
This study is a two-arm parallel randomised controlled trial comprising both outcome and cost-effectiveness analyses. A total of 244 eligible participants experiencing depressive symptoms will be randomly assigned to either the stepped care model of lifestyle-based mental health care (LSC) or the care-as-usual (CAU) at a 1:1 ratio. Participants in the LSC will access a stepped care treatment consisting of 3 steps, including self-help multicomponent LM treatment (Step 1), guided self-help based on the LM approach and low-intensity cognitive behavioural therapy for depression (Step 2), and specialist mental health services (Step 3). Participants in the CAU will be informed about their mental health condition and have unrestricted access to care. For the outcome analysis, the outcome assessments will include depressive symptoms, anxiety symptoms, insomnia symptoms, functional impairment, quality of life (QoL), health-promoting behaviours (HPBs), barriers to accessing mental health services, treatment acceptability, and treatment credibility and expectancy. For the cost-effectiveness analysis, the clinical outcome will be depressive symptoms and the economic outcome will be quality-adjusted life-years. Data will be collected at baseline, 3-month, 6-month (immediate post-treatment), 9-month follow-up, and 12-month follow-up assessements.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged 18-64 years
* Able to read and understand Cantonese
* Meeting caseness on the Patient Health Questionnaire (PHQ-9) (i.e., PHQ-9 ≥10), with symptoms persisting for four weeks of watchful waiting
* Possessing an internet-enabled iOS- or Android-operated mobile device

Exclusion Criteria:

* Meeting DSM-5 diagnosis of a severe mental illness including psychotic or bipolar disorders as determined by the Mini International Neuropsychiatric Interview 7.0.2 (MINI-7)
* Having a medical condition or neurocognitive disorder that may prevent lifestyle modifications based on the research team's clinical knowledge and experience (e.g., at high risk of fall or dietary change is not suitable as recommended by physicians or dietitians)
* Significant functional impairment as assessed by the Work and Social Adjustment Scale (WSAS) (i.e., WSAS ≥20)
* Unstable medication in the past two months
* Are receiving psychotherapy or other medical procedures (e.g., transcranial magnetic stimulation) for depression
* Current involvement in lifestyle modifications prescribed by medical (e.g., psychiatrist) or allied health professionals (e.g., clinical psychologists, dietitians)
* Prominent suicidal ideation or intent (i.e., non-fleeting intent or plan) as measured by the PHQ-9 item 9 score >2 (24-hour emergency hotlines and referral information for public mental health services will be provided)
* Participating in another clinical trial
* Pregnancy
* Hospitalisation
* Unwilling to provide informed consent or comply with the research protocol

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 244 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, 3-month, immediate post-treatment, 9-month follow-up, and 12-month follow-ups
  The PHQ-9, a 9-item questionnaire used for screening, diagnosing, and measuring the severity of depression. Participants respond to each item on a 4-point Likert-type scale ranging from 0 (not at all) to 3 (nearly every day). The total PHQ-9 score is the sum of the scores on the 9 items and ranges from 0-27. A higher score indicates more severe depressive symptoms.

SECONDARY OUTCOMES:
Change in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Baseline, immediate post-treatment, and 12-month follow-up
  The GAD-7, a 7-item questionnaire will be used to assess the severity of generalised anxiety over the past 2 weeks. Participants respond to each item on a 4-point Likert-type scale ranging from 0 (not at all) to 3 (nearly every day). The total GAD-7 score is the sum of the scores on the 7 items with a range from 0 to 21. A higher score indicates more severe generalised anxiety symptoms.
Change in the Insomnia Severity Index (ISI) | Baseline, immediate post-treatment, and 12-month follow-up
  ISI is a 7-item questionnaire that uses a 5-point Likert-type scale to measure the severity of insomnia. The total ISI score is the sum of the scores on the 7 items with a range from 0 to 28. A higher score indicates more severe insomnia symptoms.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline and immediate post-treatment
  The CEQ is a 6-item scale, with the sum of the first 3 items providing a measure of treatment credibility and the sum of the remaining 3 items examining treatment expectancy. Higher scores indicate greater credibility and success expectancy for the treatment.
Change in the Treatment Acceptability and Adherence Scale (TAAS) | Baseline and immediate post-treatment
  The TAAS a 10-item self-report questionnaire measuring on a 7-point Likert scale that extends from 1 (disagree strongly) to 7 (agree strongly). Total scores are obtained by summing across all items after negatively worded items (3, 4, 5, 7, 8, and 10) have been reverse-scored. Scores may range from 10 to 70, with higher scores indicating greater acceptability of treatment and greater anticipated ability to adhere to it.
Change in the EuroQol questionnaire (EQ-5D-5L) | Baseline, 3-month, immediate post-treatment, 9-month follow-up, and 12-month follow-ups
  The EQ-5D-5L consists of five items that measure five health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a visual analogue scale (EQ-VAS) on global health. Each health dimension has five response levels, i.e., no problems, slight, moderate, severe, and extreme problems. The EQ-5D-5L health states can be converted into a single index 'utility' score using the Hong Kong population EQ-5D-5L value set with a range of 0 (death) to 1 (perfect health) (Wong et al., 2019). The EQ-VAS ranged between 0 (worst imaginable health) and 100 (best imaginable health).
Change in the Health Promotion Lifestyle Profile II (HPLP-II) | Baseline, immediate post-treatment, and 12-month follow-up
  HPLP-II is a 52-item questionnaire scored on a 4-point Likert-type scale ranging from 1 (never) to 4 (routinely). The HPLP-II measures the overall health-promoting lifestyle and 6 subdomains of HPBs, which include health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations, and stress management. The overall health-promoting lifestyle score is the sum of the scores on the 52 items with a range from 52 to 208, whereas the score of each subdomain is the sum of the scores on the specific items (8 or 9 items) within that subdomain with a range from 8-32 or 9-36. A higher score indicates more HPBs.
Change in the Work and Social Adjustment Scale (WSAS) | Baseline, immediate post-treatment, and 12-month follow-up
  WSAS is a 5-item self-report scale that aims to evaluate impairment in function in terms of work, home management, social leisure, private leisure, and personal or family relationships (Mundt et al., 2002). The total score is the sum of the scores on the 5 items with a range from 0-40, of which 0-9 will be categorised as low impairment, 10-19 will be categorised as moderate impairment, and 20-40 will be categorised as severe impairment.
Change in the Barriers to Access to Care Evaluation Scale Version 3 (BACE) | Baseline, immediate post-treatment, and 12-month follow-up
  The BACE is a 30-item questionnaire designed to assess perceived obstacles, including practical, socioeconomic, attitudinal, and structural barriers, related to accessing mental health services. Participants respond to each item on a 4-point Likert scale from 0 (not a challenge) to 3 (a lot of challenge). The total BACE score is the sum of the 30 items with a range from 0-90. A higher score represents greater perceived barriers to receiving mental health services.
Change in the the adapted version of the Trimbos and iMTA Questionnaire for Costs associated with Psychiatric Illness (TiCP) | Baseline, 3-month, immediate post-treatment, 9-month follow-up, and 12-month follow-ups
  The TiCP is a self-report questionnaire designed to estimate the direct healthcare costs and productivity costs related to mental disorders. The TiCP assesses participants' utilisation of various healthcare services and their frequency in the past three months, which includes all types of visits to primary care (e.g., general practitioner, physiotherapist) and secondary care (e.g., medical specialist, psychologist or psychiatrist, hospital admission), medication costs, and informal care (i.e., by informal caregivers such as relatives, friends, and neighbours) they received. Additionally, information on participants' workplace absenteeism and/or reduction in productivity in paid or unpaid work due to mental health illnesses in the past month will also be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Yan-Yee Ho, PhD, Study Chair — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No